CLINICAL TRIAL: NCT02349828
Title: A Prospective, Randomized Trial of Antiviral Prophylaxis in a Population of Burn Patients
Brief Title: Antiviral Prophylaxis in a Burn Population
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI decided to stop due to divisional reorganization. No pts enrolled.
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEU-SIUSM-15-001
Record Dates: First submitted 2015-01-23; First posted 2015-01-29 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Herpes Simplex
Keywords: antiviral; herpes simplex virus; herpes; burn patients; HSV; acyclovir
MeSH Terms: conditions — Herpes Simplex | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zovirax (Active Comparator): Adult dose - 400 mg twice daily generic name: Acyclovir
  Interventions: Drug: Acyclovir
- No treatment (No Intervention): standard of care

INTERVENTIONS:
Drug: Acyclovir
  Other Names: Zovirax
  Arms: Zovirax

SUMMARY:
A prospective, randomized trial to calculate incidence of Herpes Simplex Virus in an in-patient burn population and determine efficacy of prophylactic antiviral therapy to prevent viral infection and/or reactivation. Hypothesis is that antiviral prophylaxis will be effective in reducing HSV infection/reactivation.

DETAILED DESCRIPTION:
A prospective, randomized trial of antiviral prophylaxis of at risk individuals has yet to be performed. We anticipate that the disease burden in our population of burn patients will be large, especially in patients who exhibit high risk characteristics, and hypothesize that antiviral prophylaxis will significantly reduce the incidence of Herpes Simplex Virus in the burn population. This study will have a profound impact on the treatment of burn patients both at our own institution and throughout the country. Prophylactic treatment using Acyclovir in burn patients would decrease patient morbidity, pain and suffering and would likely positively impact scarring, wound healing, and, ultimately, patient satisfaction and quality of life. Reducing the incidence of HSV infections will decrease the length of hospital stays for many patients, saving both health care expenses and resources. If prophylactic Acyclovir becomes standard of care treatment for burn patients, this treatment plan would be a tremendous public health breakthrough for preventing HSV outbreaks and could be extrapolated to researching similar protocols for other health conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Memorial Medical Center's Regional Burn Unit, both transfers and direct admissions
* Patients aged 24 months to 110 years old
* Patients presenting with thermal, flame, flash, chemical, grease or electrical burns
* Patients with second degree or higher burn to the face or burn to any part of the body of 20% TBSA or greater
* Patients, power of attorney or legally authorized representative cognitively competent to give consent.

Exclusion Criteria:

* Patients who do not wish to consent to all facets of the study
* Patients younger than 24 months
* Patients older than 110 years of age
* Patients with mechanical skin injury (ie, road rash, crush injury)
* Patients who are pregnant or become pregnant during the treatment phase of the study
* Patients with a documented allergy to Acyclovir, Famcyclovir or Valacyclovir
* Patients already taking Acyclovir, Famcyclovir or Valacyclovir
* Patients who have or develop thrombotic thrombocytopenic purpura
* Patients have or develop hemolytic uremic syndrome
* Patients concurrently taking Tizanidine, Phenytoin, Valproic Acid, Fosphenytoin, Meperidine, Micophenolic Acid, Tenofovir Disoproxil Fumarate, or Zidovudine
* Patients whom the investigator feels would be inappropriate.

Min Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
incidence of Herpes Simplex Virus | 2 weeks
  Herpes Simplex Virus 1

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Neumeister, MD, Principal Investigator — Southern Illinois Univeristy School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States